CLINICAL TRIAL: NCT05293912
Title: A Phase Ia/Ib, First-in-Human, Open-Label, Multicenter, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Efficacy of SG2501 in Subjects with Relapsed or Refractory Hematological Malignancies and Lymphoma.
Brief Title: SG2501 Safety Study in Subjects with Relapsed or Refractory Hematological Malignancies and Lymphoma.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of clinical development plan
Sponsor: Hangzhou Sumgen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSG-2501-101
Record Dates: First submitted 2022-03-01; First posted 2022-03-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hematological Malignancy; Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma | interventions — Antibodies, Bispecific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SG2501 (Experimental): SG2501 monotherapy intravenous (IV) infusion - Weekly doses
  Interventions: Drug: SG2501

INTERVENTIONS:
Drug: SG2501 — During study treatment, subjects will receive SG2501 treatment via IV infusion once every week at doses of: 0.01, 0.03, 0.1, 0.3, 1, 2, 4 and 6mg/kg.
  Other Names: Recombinant Anti-cluster of Differentiation 38(CD38)/47(CD47) Bispecific Antibody

SUMMARY:
This is a phase Ia/Ib, first-in-Human, open-Label, multicenter, dose escalation and dose expansion study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of SG2501 in subjects with relapsed or refractory hematological malignancies and lymphoma.

DETAILED DESCRIPTION:
Phase Ia will consist of two parts:an accelerated titration using single patient cohorts to evaluate SG2501 at lower dose levels(Part A), followed by dose-escalation using multipatient cohorts to establish a maximum tolerated dose(MTD)(Part B). Phase Ib will consist of dose expansion cohorts with SG2501 monotherapy in subjects with relapsed or refractory multiple myeloma(MM) or diffuse large B-cell lymphoma(DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following criteria to be eligible for participation in this study:

  1. Male or female ≥ 18 years.
  2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedurs.
  3. Cohort specific inclusion criteria.

     1. Phase Ia,dose escalation:

        • Patients with histologically or cytologically confirmed relapsed or refractory hematological malignancies and lymphoma based on WHO(2016) diagnosis who are refractory to or intolerant of established therapies known to provide clinical benefit.

        Note: the histologic subtypes that are eligible for enrollment per the 2016 WHO criteria include multiple myeloma(MM), Chronic Lymphoid Leukemias (CLL) , Waldenstrom Macroglobulinemia (WM) primary systemic amyloidosis (PSA), Hodgkin's Lymphoma(HL) and Non-Hodgkin's Lymphoma(NHL).
     2. Phase Ib, Cohort1 MM Histologically or cytologically confirmed relapsed or refractory multiple myeloma based on WHO diagnosis. Subject has received at least 3 prior anti-myeloma regimens including a proteasome inhibitor (PI), a CD38 antibody and an immunomodulatory agent.

        * Induction,bone marrow transplant with or without maintenance therapy is considered one regimen.
        * Refractory is defined as disease that is nonresponsive on therapy, or progresses within 60 days of last therapy. Nonresponsive disease is defined as either failure to achieve minimal response or development of progressive disease while on therapy
        * For subjects who received more than 1 regimen containing a PI their disease must be refractory to the most recent PI containing regimen.
        * For subiects who received more than 1 regimen containing an immunomodulatory agent their disease must be refractory to the most recent immunomodulatory agent containing regimen.
     3. Phase Ib,Cohort DLBCL

        * Histologically confirmed de novo or transformed DLBCL based on WHO diagnosis , relapsed or refractory to first line chemoimmunotherapy (eg, R-CHOP or equivalent) and second line salvage regimens or autologous hematopoetic cell transplantation, and for whom no further therapy is available that is known to provide clinical benefit.
        * Disease that is measurable or assessable for response according to Lugano Classification for lymphomas.

     Note: This may depend on the patient's mutational status, eligibility for allogeneic transplant. Patients must be willing to undergo bone marrow aspirates/biopsies per protocol specifications; These will be performed per protocol schedule to evaluate patient response to treatment.
  4. ECOG score≤ 2.
  5. Life expectancy≥ 12 weeks.
  6. Adequate hepatic function as evidenced by meeting all the following requirements:

     1. Total bilirubin≤1.5 x upper limit of normal(ULN)or≤3x ULN in patients with documented Gilbert's syndrome;
     2. Aspartate aminotransferase(AST) and alanine aminotransferase(ALT)≤2.5x ULN; AST or ALT≤5 x ULN if liver metastases are present.
  7. Renal: serum creatinine≤1.5x ULN or calculated creatinine clearance(CrCL) ≥ 50mL/min (Cockcroft-Gault Formula).
  8. Hematological function defined as:

     1. Absolute neutrophil count (ANC)≥ 10x10^9/L without growth factor support Within 7 days prior to entry;
     2. Platelet count≥75x10^9/L without transfusion within 7 days prior to entry;
     3. Hemoglobin≥ 8g/dL without transfusion within 7 days prior to entry;
     4. For leukemia: The white blood cell(WBC)count in the patient's peripheral blood must be≤20x10^9/L within 7 days of the first dose of the study drug. The patients with WBC count>20x10^9/L may be treated with hydroxyurea(maximum dose 4g/d) during the Screening period to achieve entry criteria. Hydroxyurea may be continued for the first 5 weeks of treatment(Cycle 1) to control blast counts at the discretion of the Investigator; hydroxyurea must be stopped after the first 5 weeks of treatment. For these patients where is not absolute lower level for neutrophils or platelets for enrollment Platelets and RBCcan be transfused as clinically indicated. Hematopoietic growth factors are prohibited.
  9. Coagulation tests INR≤ 2 or prothrombin time ≤ 2×ULN.
  10. Baseline Left Ventricular Ejection Fraction (LVEF) ≥ 50% measured by multiple-gated acquisition (MUGA) or echocardiogram (ECHO) or lower limit for institutional normal value.
  11. Recovery, to Grade 0-1, from adverse events related to prior anticancer therapy except alopecia, Grade ≤2 sensory neuropathy, lymphopenia, and endocrinopathies controlled with hormone replacement therapy.
  12. Archival tumor tissue will be requested from all patients for exploratory biomarker research. If archival tumor tissue is not available, a fresh biopsy, taken from a readily accessible tumor lesion will be obtained. A patient who does not have a readily accessible tumor may still be enrolled. Tumor tissue is not required for enrollment however an official pathology report documenting the patient's cancer will be required.
  13. Patients must be willing to undergo transfusion with RBCs and/or platelets if clinically indicated.
  14. Subjects (women of child-bearing potential and males with fertile female partner) must be willing to use currently accepted reliable contraception method throughout the treatment period and for at least three months following the last dose of study drug. These measures include, but are not limited to, oral or implantable injections of hormonal contraceptives; intrauterine birth control ring or placement of IUS intrauterine device); or use of barrier methods such as condoms or septum and spermicide products. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Women of childbearing age must have a negative pregnancy test.

Exclusion Criteria:

* Patients who meet any of the following criteria cannot be enrolled:

  1. Symptomatic central nervous system (CNS) metastases or leptomeningeal disease or primary CNS tumors. Patients with asymptomatic CNS metastases who are radiologically and neurologically stable ≥ 4 weeks following CNS-directed therapy and are off steroids for at least 2 weeks prior to dosing may be eligible for study entry.
  2. For lymphoma: red blood cell transfusion within 2 weeks prior to study entry.
  3. History of hemolytic anemia of any cause (including Evans syndrome) within 3 months.
  4. Positive direct antiglobulin test (DAT).
  5. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months, serious arrhythmias requiring medication.
  6. Significant (requiring anticoagulation or transfusion) thrombotic or hemorrhagic event within 6 months prior to study entry.
  7. Active infection requiring intravenous therapy within 2 weeks prior to study drug administration.
  8. HIV infection with a current or a history of AIDS-defining illness or HIV infection with a CD4+ T cell count < 350 cells/μL regardless of history of AIDS-defining illness.
  9. Patients with active viral (any etiology) hepatitis are excluded. Patients with serologic evidence of chronic HBV infection (defined by a positive hepatitis B surface antigen test and a positive anti-hepatitis core antibody test) who have a viral load below the limit quantification (HBV DNA titer < 200 IU/mL) and are not currently on viral suppressive therapy may be eligible and should be discussed with the Medical Monitor. Patients with a history of HCV infection should have completed curative antiviral treatment and have a viral load below the limit of quantification.
  10. Anticancer therapy within 5 half-lives or 4 weeks (whichever is shorter) or radiation therapy within 14 days prior to study entry; palliative radiotherapy to a single area of metastasis within 2 weeks prior to study entry. If a patient is receiving high dose cytarabine, liposomal cytarabine, or standard-dose cytarabine (100-200 mg/m2/day), the patient must be off the drug for at least 2 weeks or until the patient has recovered from toxic effects.
  11. Previous exposure to any anti-CD47 monoclonal antibody or SIRPα antibody or SIRPα fusion construct.
  12. Major surgery within 4 weeks prior to study entry.
  13. Allergy to study drug or components of its formulation or history of a Grade 3-4 allergic reaction to treatment with another protein product.
  14. Pregnant or breast-feeding females.
  15. Men with a partner of childbearing potential who do not consent to use two acceptable methods of birth control during treatment and for an additional 90 days after the last administration of study drug.
  16. Prior or concurrent malignancy within 2 years prior to entry, other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, superficial bladder cancer, or prostate cancer under active surveillance.
  17. Concomitant active autoimmune disease or history of autoimmune disease requiring systemic treatment within 2 years prior to study entry except vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus or hypothyroidism which can be managed by replacement therapy.
  18. Known active tuberculosis.
  19. Known active SARS-CoV-2 infection.
  20. Use of systemic corticosteroids in a dose equivalent to > 10 mg/d of prednisone or other immunosuppressive agent within 2 weeks prior to entry; Use of inhaled, topical, or ophthalmological steroids are allowed. Short term use of corticosteroids at doses equivalent to > 10 mg/d of prednisone (e.g., pre-medication for IV contrast) is allowed.
  21. Received allogeneic stem cell transplantation within 3 months prior to entry, or GVHD after allogeneic stem cell transplantation requiring systemic immunosuppressants, such as cyclosporin or tacrolimus.
  22. Symptomatic intrinsic lung disease (chronic obstructive pulmonary disease, pulmonary fibrosis).
  23. Live virus vaccine within 28 days prior to study entry.
  24. Allergy to study drug or components of its formulation or history of a Grade 3-4 allergic reaction to treatment with another protein product.
  25. Intolerant to IV infusion.
  26. Any other serious underlying medical (e.g. uncontrolled diabetes mellitus, uncontrolled hypertension, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.
  27. Any condition that the Investigator or primary physician believes may not be appropriate for participating the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with AEs and SAEs | At the end of treatment phase (24 weeks)
  To evaluate the safety and tolerability of SG2501 [Adverse events (AEs), Serious Adverse Events (SAE)].
The Maximum tolerated dose (MTD) and Recommended Phase 2 dose (RP2D) for SG2501 | At the end of treatment phase (24 weeks)
  MTD/Recommended Phase 2 dose (RP2D) determined by DLTs and other safety data,as well as available PK data.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): AUC | At the end of treatment phase (24 weeks)
  The area under the curve (AUC) of serum concentration of the drug after the administration.
Pharmacokinetics (PK): Cmax | At the end of treatment phase (24 weeks)
  Maximum Concentration (Cmax) of the drug after administration.
Immunogenicity: percentage of ADA positive patients | At the end of treatment phase (24 weeks)
  Number and percentage of subjects with ADAs.
Preliminary anti-tumor activity of SG2501 (Objective Response Rate) | At the end of treatment phase (24 weeks)
  To assess the preliminary antitumor activity of SG2501 following IV infusion in subjects with relapsed or refractory hematological malignancies and lymphoma.
Receptor occupancy | At the end of treatment phase (24 weeks)
  CD47 and CD38 receptor occupancy (%).
Immune-cell type assessment | At the end of treatment phase (24 weeks)
  Cell counts and percentages of T lymphocytes, NK cells, and B lymphocytes, including but not limited to CD4+, CD8+ T lymphocytes, CD38+MDSCs, CD38+Tregs, CD38+Bregs, CD16+CD56+, CD16+CD56dim assessed by FACS analysis of peripheral blood leukocytes.
Cytokine level | At the end of treatment phase (24 weeks)
  Levels of inflammatory cytokine biomarkers, including, but not limited to TNF α, IFN γ, IL-2, IL-4, IL-6, IL-8 and IL-1β.
Correlation antitumor activity | At the end of treatment phase (24 weeks)
  To explore the correlation of SG2501 antitumor activity and potential tumor markers, including but not limited to CD47and CD38 expression in archived tumor samples.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Northside Hospital, Atlanta, Georgia
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Westchester Medical Center, Hawthorne, New York
  - Novant Health Forsyth Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Novant Health Cancer Institute Hematology - Forsyth, Winston-Salem, North Carolina
  - Gabrail Cancer Center Research, LLC, Canton, Ohio
  - Texas Oncology / Baylor Charles A. Sammons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No